CLINICAL TRIAL: NCT04132115
Title: Prospective Study Evaluating Plasma Exposure of Optimized Antibiotic Therapy According to TDM in Patients With Subarachnoid Haemorrhage (ES) and Cerebral Haemorrhage (EC)
Brief Title: Optimized Antibiotic Therapy in Patients With Subarachnoid Haemorrhage (ES) and Cerebral Haemorrhage (EC)
Acronym: TANDEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Luigi Vetrugno, Clinical Professor, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: CEUR-2019-Os-162
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Therapeutic Drug Monitoring; Subarachnoid Hemorrhage; Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Subarachnoid Hemorrhage; Therapeutic Drug Monitoring
MeSH Terms: conditions — Subarachnoid Hemorrhage; Cerebral Hemorrhage | interventions — Piperacillin, Tazobactam Drug Combination; Meropenem; Daptomycin; ceftobiprole; Linezolid; Vancomycin; Fluconazole; Acyclovir; Gentamicins; Amikacin; Ganciclovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Piperacillin/tazobactam — Therapeutic drug monitoring (TDM) of this antibiotic plasma concentration
Drug: Meropenem — Therapeutic drug monitoring (TDM) of this antibiotic plasma concentration
Drug: Daptomycin — Therapeutic drug monitoring (TDM) of this antibiotic plasma concentration
Drug: Ceftobiprole — Therapeutic drug monitoring (TDM) of this antibiotic plasma concentration
Drug: Linezolid — Therapeutic drug monitoring (TDM) of this antibiotic plasma concentration
Drug: Vancomycin — Therapeutic drug monitoring(TDM) of this antibiotic plasma concentration
Drug: Fluconazol — Therapeutic drug monitoring (TDM) of this antifungal plasma concentration
Drug: Acyclovir — Therapeutic drug monitoring (TDM) of this antiviral plasma concentration
Drug: Gentamicins — Therapeutic drug monitoring (TDM) of this antibiotic plasma concentration
Drug: Amikacin — Therapeutic drug monitoring (TDM) of this antibiotic plasma concentration
Drug: Ganciclovir — Therapeutic drug monitoring (TDM) of this antiviral plasma concentration

SUMMARY:
A recent prospective observational clinical study conducted in an intensive care unit of a third level US university hospital showed that 94% of patients with ES and 50% of those with EC had an ARC for a duration of at least one day during the hospital stay.

Although there is currently a great deal of evidence describing ARC in various subgroups of critically ill patients, on the other hand there is little documentation regarding the effect that ARC can have on exposure to renally eliminated drugs.

Therefore, the aim of this study is to prospectively evaluate the proportion of plasma under-exposure to hydrophilic antimicrobials in patients with ES or EC and with ARC, in order to verify whether the recommended dosage regimens for these drugs are adequate for reaching the pharmacodynamic targets of therapeutic efficacy.

DETAILED DESCRIPTION:
Haemorrhagic stroke is a devastating disease with a high rate of disability and mortality. In addition to the direct effects of the haemorrhagic event and to the secondary neurological complications, patients with haemorrhagic strokes are predisposed to medical complications that can have a direct impact on both clinical outcome and treatment costs. It has been estimated that between 79% and 100% of patients with subarachnoid haemorrhage (ES) and cerebral haemorrhage (EC) have at least one of these complications. Among them, the most common are infections, seizures, hyponatremia, hypomagnesemia, hypokalemia and venous thromboembolism.

A possible reason that can be responsible for such a high frequency of complications, especially infectious, can be identified in a pathophysiological alteration of the circulatory and renal haemodynamics of this population. Specifically, these patients frequently have a hyperdynamic state which results in a high renal clearance (CrCl) (augmented renal clearance - ARC, defined as a measured CrCl ≥ 130 ml/min/1.73m2). In this regard, a recent prospective observational clinical study conducted in an intensive care unit of a third level US university hospital showed that 94% of patients with ES and 50% of those with EC had an ARC for a duration of at least one day during the hospital stay.

In consideration of the fact that the ARC has been historically underestimated and that an accurate assessment of renal function through the measured CrCl is not regularly carried out on all patients even if they are critical, the main risk from the point of view of therapeutic appropriateness is that of not adjust the dosing regimen of drugs eliminated through the kidney in relation to the presence and extent of the ARC. Moreover, the clinician often ignores the time course of the ARC as well as the modalities with which to carry out the dosage adjustment. This could lead to sub-therapeutic concentrations for renally excreted drugs, as typically are water-soluble antibiotics such as beta-lactams, aminoglycosides, daptomycin, linezolid, antifungal fluconazole and antivirals ganciclovir and aciclovir, resulting in an increase in the risk of therapeutic failure.

Although there is currently a great deal of evidence describing ARC in various subgroups of critically ill patients, on the other hand there is little documentation regarding the effect that ARC can have on exposure to renally eliminated drugs.

Therefore, the aim of this study is to prospectively evaluate the proportion of plasma under-exposure to hydrophilic antimicrobials in patients with ES or EC and with ARC, in order to verify whether the recommended dosage regimens for these drugs are adequate for reaching the pharmacodynamic targets of therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes > 18 years admitted for ES or EC
* Patients to which one or more water-soluble antibiotics, antifungals or antivirals subject of the present study are prescribed
* Patients who present ARC

Exclusion Criteria:

* Patients in whom the plasma samples are contaminated
* Patients in whom the plasma samples are performed in a way that does not comply with the prepared company protocol.
* Patients with BMI < 18 kg / m2.
* Patients with a serum creatinine > 1.4 mg / dL at entry
* Pregnant patients.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU due to intracranial haemorrage or subaracnoid haemorrage
Sampling Method: Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Underexposure to antimicrobial therapy | 2 years from the date of approval
  Prospective evaluation of the proportion of plasma underexposure to hydrophilic antimicrobials due to ARC in patients with subarachnoid haemorrhage (ES) and / or cerebral haemorrhage (EC).

SECONDARY OUTCOMES:
T > MIC | 2 years from the date of approval
  Evaluation of the achievement of the pharmacokinetic / pharmacodynamic target of therapeutic efficacy through the calculation of the parameter T > MIC
AUC / MIC | 2 years from the date of approval
  Evaluation of the achievement of the pharmacokinetic / pharmacodynamic target of therapeutic efficacy through the calculation of the parameter AUC / MIC
Performance of ClCr estimation formulas | 2 years from the date of approval
  Evaluation of the performance of the common CrCl estimation formulas compared to the CrCl measured in the estimation of the systemic clearance of the drugs being studied

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Anesthesiology and Intensive Care Clinic - Department of Medicine - ASUIUD, Udine
  - Terapia Intensiva 1, Udine

IPD SHARING:
Plan to Share IPD: Yes
Database will be available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code